CLINICAL TRIAL: NCT06659029
Title: PRIMULA Preg (Prospective Registry Investigating Maternal and Infant Outcomes in Anifrolumab Users): The AstraZeneca Pregnancy Study for Anifrolumab
Brief Title: Prospective Registry Investigating Maternal and Infant Outcomes in Anifrolumab Users
Acronym: PRIMULA_Preg
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00051
Record Dates: First submitted 2024-10-14; First posted 2024-10-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Chronic autoimmune disease; Immunosuppressants; Corticosteroids; Human monoclonal antibody (IgG1ƙ mAb); Post Marketing Requirements (PMR) study; Pregnancy; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed cohort: Pregnant individuals with a diagnosis of moderate/severe SLE who are exposed to anifrolumab at any time during pregnancy
  Interventions: Drug: Anifrolumab
- Unexposed cohort: Pregnant individuals with a diagnosis of moderate/severe SLE who are not exposed to anifrolumab at any time during pregnancy but who are exposed to other products for the treatment of SLE

INTERVENTIONS:
Drug: Anifrolumab — Anifrolumab is a human monoclonal antibody that binds to subunit 1 of the type 1 interferon receptor, which was developed based on the evidence supporting the role of type 1 interferon pathway in SLE. Clinical trial evidence from TULIP 1 and TULIP 2 have showed that monthly intravenous administration of anifrolumab led to a higher percentage of patients with a response, assessed with the British Isles Lupus Assessment Group-based Composite Lupus Assessment, compared with patients receiving placebo. Moreover, the phase II MUSE study showed that administration of anifrolumab resulted in substantially reduce disease activity, as measured by the SLE Responder Index, compared to patients receiving placebo. Anifrolumab was approved by the FDA and EMA in July 2021 and February 2022, respectively, for the treatment of adult patients with moderate to severe SLE who are receiving standard therapy.
  Other Names: Saphnelo
  Groups: Exposed cohort

SUMMARY:
PRIMULA Preg (Prospective Registry Investigating Maternal and Infant Outcomes in Anifrolumab Users) is a prospective, observational cohort study designed to evaluate the association between anifrolumab exposure during pregnancy and subsequent adverse maternal, fetal, and infant outcomes. This study will fulfil an FDA post-marketing requirement.

DETAILED DESCRIPTION:
PRIMULA Preg (Prospective Registry Investigating Maternal and Infant Outcomes in Anifrolumab Users) is a US-based, prospective, observational cohort study designed to evaluate the association between anifrolumab exposure during pregnancy and subsequent adverse maternal, fetal, and infant outcomes. The objective of the pregnancy registry is to compare adverse maternal, fetal, and infant outcomes of pregnant individuals with moderate/severe systemic lupus erythematosus (SLE) who are exposed to anifrolumab during pregnancy with outcomes in an internal comparison cohort of pregnant individuals with moderate/severe SLE who are not exposed to anifrolumab during pregnancy. Participation in the registry is voluntary and participants can withdraw their consent to participate at any time. The study is strictly observational; the schedule of office visits and all treatment regimens will be determined by HCPs. Only data that are documented in patients' medical records during medical care will be actively collected. No additional laboratory tests or HCP assessments will be required as part of this registry. This study will fulfil an FDA post-marketing requirement.

ELIGIBILITY:
Inclusion Criteria:

Exposed cohort

1. Currently or recently (within 1 year of pregnancy outcome) pregnant
2. Diagnosis of moderate/severe SLE
3. Consent to participate
4. Authorization for their HCP(s) to provide data to the registry
5. Exposure to at least 1 dose of anifrolumab at any time during pregnancy

Unexposed cohort

1. Currently or recently pregnant
2. Diagnosis of moderate/severe SLE
3. Consent to participate
4. Authorization for their HCP(s) to provide data to the registry
5. Exposure to other products for the treatment of moderate/severe SLE

Exclusion Criteria:

Exposed cohort

1. Occurrence of pregnancy outcome prior to first contact (for enrollment) with the Virtual Research Coordination Center (retrospectively enrolled)
2. Exposure to known teratogens and/or investigational medications during pregnancy

Unexposed cohort

1. Occurrence of pregnancy outcome prior to first contact with the Virtual Research Coordination Center (retrospectively enrolled)
2. Exposure to known teratogens and/or investigational medications during pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include 2 cohorts of pregnant individuals: a cohort of individuals with moderate/severe SLE who are exposed to anifrolumab and a cohort of individuals with moderate/severe SLE who are unexposed to anifrolumab but who are exposed to other products for the treatment of SLE.
Sampling Method: Non-Probability Sample
Enrollment: 442 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2031-04-15 (Estimated); Study Completion 2031-04-15 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of all major congenital malformations (MCMs) | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  An abnormality of body structure or function that is present at birth, is of prenatal origin (i.e., birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention. Relevant exposure window is limited to 1st trimester of pregnancy.

SECONDARY OUTCOMES:
Composite outcome of all minor congenital malformations | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  An anomaly or abnormality of body structure that is present at birth, is of prenatal origin (i.e., birth defect), poses no significant health problem in the neonatal period, and tends to have limited social or cosmetic consequences for the affected individual. Relevant exposure window includes any trimester of pregnancy.
Worsening of underlying disease | From date of conception (DOC) to pregnancy outcome, up to 42 weeks of pregnancy
  Any increase in disease activity or severity in the pregnancy period compared to the baseline period (6 months prior to pregnancy) as assessed by the disease flare or disease activity algorithms or as reported by an HCP. Relevant exposure window includes any trimester of pregnancy.
Premature rupture of membranes | From date of conception (DOC) to pregnancy outcome, up to 42 weeks of pregnancy
  A disorder of pregnancy defined as rupture of membranes before the onset of labor. Relevant exposure window includes any trimester of pregnancy.
Pregnancy-induced hypertension | From 20 gestational weeks to pregnancy outcome, up to 42 weeks of pregnancy
  A disorder of pregnancy defined as a systolic blood pressure 140 mmHg or more or a diastolic blood pressure of 90 mmHg or more, or both, on 2 occasions at least 4 hours apart after 20 weeks gestation, in a woman with a previously normal blood pressure. Relevant exposure window includes any trimester of pregnancy.
Composite outcome of preeclampsia/eclampsia | From 20 gestational weeks to pregnancy outcome, up to 42 weeks of pregnancy
  Preeclampsia is a disorder of pregnancy associated with new-onset hypertension, which occurs most often after 20 weeks of gestation and frequently near term, and proteinuria. Or, in the absence of proteinuria, it is defined as new-onset hypertension with the new onset of any of the following:
  * Thrombocytopenia: platelet count less <100 ,000/mL
  * Renal insufficiency: serum creatinine concentrations >1.1mg/dL or a doubling of the serum creatinine concentration in the absence of other renal disease
  * Impaired liver function: elevated blood concentrations of liver transaminases to twice normal concentration
  * Pulmonary edema
  * New-onset headache unresponsive to medication and not accounted for by alternative diagnoses or visual symptoms.
  Eclampsia is new-onset tonic-clonic, focal, or multifocal seizures in the absence of other causative conditions such as epilepsy, cerebral arterial ischemia and infarction, intracranial hemorrhage, or drug use.
Maternal hospitalization for serious illness | From date of conception (DOC) to pregnancy outcome, up to 42 weeks of pregnancy
  An inpatient hospital admission unrelated to delivery occurring during pregnancy. Relevant exposure window includes any trimester of pregnancy.
Spontaneous abortion | From date of conception (DOC) to <20 gestational weeks
  An involuntary fetal loss or the expulsion of the products of conception occurring at <20 gestational weeks.
Elective termination | From date of conception (DOC) to pregnancy outcome, up to 24 weeks of pregnancy
  An intervention that is intended to terminate a suspected or known ongoing intrauterine pregnancy and that does not result in a live birth. Relevant exposure window includes any trimester of pregnancy.
Emergency caesarean section | From date of conception (DOC) to pregnancy outcome, up to 42 weeks of pregnancy
  A cesarean delivery that is performed due an immediate threat to the health or safety of the fetus and/or the mother. Relevant exposure window includes any trimester of pregnancy.
Preterm birth | From date of conception (DOC) up to 37 gestational weeks
  A live birth occurring at <37 gestational weeks.
Small for gestational age | At delivery of live birth
  Birthweight <10th percentile for sex and gestational age using standard growth charts for full and preterm live-born infants. Relevant exposure window includes any trimester of pregnancy.
Postnatal growth deficiency | At 4 and 12 months of infant age
  Weight, length, or head circumference in <10th percentile for sex and chronological age using standard growth charts. Relevant exposure window includes any trimester of pregnancy.
Infant developmental delay | At 4 and 12 months of infant age
  Failure to achieve the developmental milestones for chronological age, as defined by the CDC. Relevant exposure window includes any trimester of pregnancy.
Infant hospitalization for serious illness | From birth to 1 year of infant age
  An inpatient hospital admission occurring in the first year of life. Relevant exposure window includes any trimester of pregnancy.
Infant serious or opportunistic infection | From birth to 1 year of infant age
  An infection that occurs within an infant's first year of life and is either opportunistic (i.e., occurs more often or is more severe in people with weakened immune systems than in people with healthy immune systems) or serious (i.e., results in significant disability, incapacity, or death; is life-threatening; requires inpatient or prolonged hospitalization; or is considered medically important). Relevant exposure window includes any trimester of pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of Companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ will accept requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of IPD sharing timelines, please refer to AZ disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the anonymized individual patient-level data via a secure research environment Vivli.org. A signed data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/